CLINICAL TRIAL: NCT07158424
Title: Effects of Serious Games on Cognitive Function, Balance, and Quality of Life in Children With Cerebral Palsy: a Randomized Controlled Trial
Brief Title: Serious Games for Serious Outcomes: Enhancing Cognition, Balance, and Quality of Life in Children With Cerebral Palsy
Acronym: Games4CP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nataliya Hrabarchuk (Industry)
Collaborators: Hasselt University (Other)
Responsible Party: Sponsor-Investigator, Nataliya Hrabarchuk, Dr., Elita Rehabilitation Center
Organization: Elita Rehabilitation Center (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ElitaRehab
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard rehabilitation program + serious games (Experimental): Participants in the experimental groups engage in daily sessions of serious games from the Vana Vital Platform. Each child play for 30 minutes per day over 10 training days.
  In addition, participants continue their intensive rehabilitation program.
  Interventions: Procedure: Serious games; Procedure: Intensive rehabilitation
- Standard rehabilitation program + 30 extra minutes of physical therapy (Active Comparator): Participants receive their intensive rehabilitation program, with an additional 30 minutes of physical therapy
  Interventions: Procedure: Intensive rehabilitation; Procedure: Physical therapy
- Standard rehabilitation program only (Active Comparator): Participants receive their intensive rehabilitation program.
  Interventions: Procedure: Intensive rehabilitation

INTERVENTIONS:
Procedure: Serious games — Participants in the experimental groups engage in daily sessions of serious games from the Vana Vital Platform (Super Surfer, Hungry Woo, Paddle Waddle, Woo's Wonderful World Adventure). Each child will for 30 minutes per day over 10 training days.
  Arms: Standard rehabilitation program + serious games
Procedure: Intensive rehabilitation — Participants receive their intensive rehabilitation program, which includes:
  30 minutes of physical therapy (PT) 20 minutes of occupational therapy 5 minutes of spinal manipulative therapy 60 minutes of full-body massage with reflexotherapy 15 minutes of joint mobilization 15 minutes of treadmill gait training (with or without suspension) 15 minutes of strength training 30 minutes of group rhythmic gymnastics
Procedure: Physical therapy — Participants receive an additional 30 minutes of physical therapy (PT)
  Arms: Standard rehabilitation program + 30 extra minutes of physical therapy

SUMMARY:
Children with cerebral palsy (CP) often face challenges with balance, movement, and skills such as memory, problem-solving, and attention. These difficulties can affect not only daily activities but also their quality of life. Rehabilitation usually focuses on physical therapy, but recent research shows that combining movement training with cognitive tasks may be even more effective.

What we are studying. This study is focused at whether serious games from the Vana Vital platform-that was specifically designed for rehabilitation-can improve balance, cognition, and quality of life in children with CP. These games are not ordinary video games: they were created to encourage children to move, focus, and solve problems at the same time (dual-tasking).

The expected benefits include:

* Better trunk control and stability.
* Improved memory, attention, and reasoning.
* Enhanced participation in daily life and overall well-being.

Takeaway. This study is exploring an innovative approach to rehabilitation: using technology and games not only to strengthen the body but also to train the mind. If successful, this method may provide a fun, effective, and family-friendly addition to traditional therapies for children with CP.

DETAILED DESCRIPTION:
Background. Cerebral palsy (CP) is one of the most common causes of movement difficulties in children. It is a lifelong condition that affects posture, coordination, and the ability to control movements. Many children with CP also experience challenges in other areas, such as attention, memory, and problem-solving. These challenges can make everyday tasks, school activities, and social participation more difficult.

Traditional rehabilitation programs focus on improving physical functions, especially motor control and balance. Training only movement may not be enough. Children may benefit from approaches that combine movement and cognitive training-practicing how to move while also thinking, remembering, or making quick decisions.

This idea is called dual-tasking: doing two things at the same time, such as walking while answering a question, or maintaining balance while remembering a sequence. In real life, dual-tasking is what we do constantly-walking while talking to a friend, keeping balance while carrying a schoolbag, or focusing in class while sitting upright. For children with CP, dual-tasking can be particularly difficult, but also particularly beneficial to practice.

Serious games are a new, innovative way to provide this training. Unlike ordinary video games, serious games are designed specifically for therapeutic purposes. They are meant to be engaging and motivating for children, while at the same time targeting key skills in motor and cognitive development.

What Makes This Study Unique. This study is among the first randomized controlled trials to test the Vana Vital platform-a suite of computer-based serious games that combine physical movements with cognitive tasks. Instead of repetitive exercises, children engage in playful adventures that require them to move their bodies while also solving challenges.

Study Design in Practice. The study follows the structure of a prospective, single-blind randomized controlled trial, which means that children are randomly assigned to groups, and the evaluators do not know which group each child belongs to (to reduce bias).

Group allocation:

Experimental Group 1: Standard rehabilitation program + serious games. Control Group 1: Standard rehabilitation program only. Control Group 2: Standard program + 30 extra minutes of physical therapy daily.

This design allows researchers to see whether serious games add benefits beyond standard care.

Expected outcomes for children include:

Stronger trunk control and better stability when sitting, standing, or walking. Improved memory, attention, and problem-solving skills. A more positive experience of rehabilitation, making therapy feel less like work and more like play.

Potential improvements in everyday life, such as sitting upright in school, playing with peers, or participating in family activities.

What Health Care Providers Can Expect For clinicians, this study provides structured evidence on the feasibility and effectiveness of adding game-based dual-task training to rehabilitation.

Conclusion This study represents a step forward in child-centered rehabilitation. Instead of seeing therapy as hard work, children can experience it as an adventure with Woo in fun, interactive worlds. By training both the body and the mind, serious games have the potential to improve balance, cognition, and overall quality of life for children with cerebral palsy.

The results of this randomized controlled trial will help healthcare providers understand whether game-based dual-tasking should become a regular part of rehabilitation programs-and will give families hope for more enjoyable, effective, and innovative ways to support their children's development.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral palsy
* Ability to attend the educational institutions
* GMFCS I, II, III

Exclusion Criteria:

* GMFCS IV, V
* Uncooperative behaviour
* Uncontrolled seizures

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-01-02 (Estimated); Study Completion 2026-01-02 (Estimated)

PRIMARY OUTCOMES:
Score of the Trunk control measurement scale (TCMS) | Baseline and 2 weeks
  The TCMS is a standardized test used to evaluate trunk control in children with cerebral palsy. Trunk control is essential for posture, balance, and movement. A physiotherapist administers the test while the child sits without back or arm support and performs tasks that assess static sitting, selective trunk movements, and dynamic reaching. Each task is scored from 0 (unable) to 2 (able), with a maximum total of 58 points: 20 for static sitting, 28 for selective movement, and 10 for dynamic reaching. Higher scores indicate better trunk control and postural stability. Lower scores reflect greater difficulty with maintaining balance and controlling trunk movements. The test usually takes 15-20 minutes to complete and has been validated for children with CP. Changes in TCMS scores are considered clinically meaningful, as they reflect improvements in motor function, daily activities, and participation.

SECONDARY OUTCOMES:
Characteristics of the Static Balance Test | Baseline and 2 weeks
  The Static Balance Test is a computerized assessment delivered through the Vana Vital platform to measure a child's ability to maintain a steady posture while standing still. During the test, the child stands on a Nintendo Wii balance board, and subtle movements of the body are recorded by sensors. The system quantifies postural sway in multiple directions (forward-backward, left-right) and provides objective data on trunk and overall balance control. The test is performed under standardized conditions, lasting 30 seconds overall per trial, with the child instructed to stand as still as possible. Results are expressed as stability scores. Lower sway values reflect better postural stability, while higher sway values indicate reduced balance control. The test is non-invasive, quick to administer, and was specifically designed for children with cerebral palsy. Improvements over time are interpreted as gains in trunk stability and postural control.
Score of the cognitive tests from Sway Medical platform | Baseline and 2 weeks
  The SWAY Medical platform provides sensor-based cognitive assessments designed for use on a tablet or smartphone. In this study, children complete short interactive tasks that measure key aspects of cognitive function, including executive functions, attention, and working memory. The tests are administered through a touch screen, requiring children to respond quickly and accurately to visual or auditory prompts. Each task lasts up to 5 mins, has 3 attempts, and provides objective, quantitative scores. The assessments are non-invasive, and validated for use in pediatric and rehabilitation settings. Results allow clinicians to monitor changes in cognition alongside motor outcomes, helping to evaluate the added value of dual-task serious game interventions in children with cerebral palsy.
Score of the RAVEN's coloured progressive matrices (RCMP) | Baseline and 2 weeks
  The RCPM is a non-verbal cognitive assessment used in children to measure general intelligence, focusing on reasoning and abstract thinking. It consists of a series of visual patterns with one piece missing; the child is asked to choose the correct missing piece from several options. The coloured version is specifically designed for younger children and those with developmental or physical challenges, as the coloured backgrounds help sustain attention and motivation. The test requires no reading, writing, or spoken language, making it suitable for children with CP and varying communication abilities. Administration typically takes 15-20 minutes. Scores are reported as the total number of correct responses (0-36), with higher scores reflecting stronger general intelligence. Results are often compared to age-based normative data to determine developmental level. The RCPM is quick, reliable, and sensitive to cognitive changes in clinical and rehabilitation research.
Score of the Pediatric Quality of Life Enjoyment and Satisfaction Questionnaire (PQ-LES-Q) | Baseline and 2 weeks
  The PQ-LES-Q is a brief, standardized questionnaire used to assess short-term changes in quality of life in children and adolescents. It evaluates domains such as physical health, mood, school performance, social relationships, and overall life satisfaction. Each item is scored on a Likert-type scale (1 = Strongly Disagree to 5 = Strongly Agree), with higher total scores reflecting greater quality of life and satisfaction. The measure is child-friendly, quick to administer (approximately 5-10 minutes), and sensitive to short-term improvements during rehabilitation programs. It complements objective motor and cognitive outcomes by capturing how children feel and function in everyday life, thereby providing a holistic picture of the impact of serious game-based interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Elita Rehabilitation Center, Lviv, Lviv Oblast, Ukraine

IPD SHARING:
Plan to Share IPD: No
This study involves children with cerebral palsy, who are considered a vulnerable population. Informed consent procedures clearly state that individual-level data will not be shared and that all personal information will remain coded and confidential. Therefore, no individual participant data (IPD) will be made publicly available. Only aggregated, de-identified results will be reported in scientific publications and presentations.

REFERENCES:
- [Background] Endicott J, Nee J, Yang R, Wohlberg C. Pediatric Quality of Life Enjoyment and Satisfaction Questionnaire (PQ-LES-Q): reliability and validity. J Am Acad Child Adolesc Psychiatry. 2006 Apr;45(4):401-7. doi: 10.1097/01.chi.0000198590.38325.81. PMID 16601644
- [Background] Pueyo R, Junque C, Vendrell P, Narberhaus A, Segarra D. Raven's Coloured Progressive Matrices as a measure of cognitive functioning in Cerebral Palsy. J Intellect Disabil Res. 2008 May;52(Pt 5):437-45. doi: 10.1111/j.1365-2788.2008.01045.x. Epub 2008 Feb 28. PMID 18312310
- [Background] Heyrman L, Molenaers G, Desloovere K, Verheyden G, De Cat J, Monbaliu E, Feys H. A clinical tool to measure trunk control in children with cerebral palsy: the Trunk Control Measurement Scale. Res Dev Disabil. 2011 Nov-Dec;32(6):2624-35. doi: 10.1016/j.ridd.2011.06.012. Epub 2011 Jul 14. PMID 21757321
- [Background] Kushnir A, Kachmar O. Intensive Neurophysiological Rehabilitation System for children with cerebral palsy: a quasi-randomized controlled trial. BMC Neurol. 2023 Apr 20;23(1):157. doi: 10.1186/s12883-023-03216-4. PMID 37081406
- [Background] Kachmar O, Kushnir A, Fedchyshyn B, Cristiano J, O'Flaherty J, Helland K, Johnson G, Puig D. Personalized balance games for children with cerebral palsy: A pilot study. J Pediatr Rehabil Med. 2021;14(2):237-245. doi: 10.3233/PRM-190666. PMID 33720857
- [Background] Szturm T, Parmar ST, Mehta K, Shetty DR, Kanitkar A, Eskicioglu R, Gaonkar N. Game-Based Dual-Task Exercise Program for Children with Cerebral Palsy: Blending Balance, Visuomotor and Cognitive Training: Feasibility Randomized Control Trial. Sensors (Basel). 2022 Jan 19;22(3):761. doi: 10.3390/s22030761. PMID 35161508
- [Background] Stadskleiv K. Cognitive functioning in children with cerebral palsy. Dev Med Child Neurol. 2020 Mar;62(3):283-289. doi: 10.1111/dmcn.14463. Epub 2020 Jan 9. PMID 32010976
- See also: Vana Vital platform that collects the serious games that are used in the study — https://vanavital.com
- See also: Sway Medical platform that contains tests to assess cognition — https://www.swaymedical.com